CLINICAL TRIAL: NCT01121731
Title: Phase I/II, Multicenter, Randomized, Open,Active-Controlled, ClinicalTrial to Evaluate PK, PD, Safety and Tolerability Of Interferon Alfa 5, S.C. 3 Times Per Week, For 29 Days, To Treat-Experienced Pat. With Genotype-1 Chronic Hepatitis C
Brief Title: A Phase I/II Clinical Trial With Interferon Alfa 5 in Treatment-Experienced Patients With Genotype-1 Chronic Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Digna Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAHE001-CHC-01; 2009-012924-10 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Hepatitis C Virus Infection; Genotype 1; Treatment-Experienced Patients; Relapses
Keywords: Chronic Hepatitis C Viral Infection; Interferon alfa-5; Interferon
MeSH Terms: conditions — Recurrence | interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interferon α-5 (Experimental)
  Interventions: Drug: Interferon α-5
- Interferon α-5 plus Interferon α-2b (Experimental)
  Interventions: Drug: Interferon-α5 plus Interferon-α 2b
- Interferon α-2b (INTRON® A) (Active Comparator)
  Interventions: Drug: Interferon α-2b (INTRON® A)

INTERVENTIONS:
Drug: Interferon α-5 — 3 MIU or safe dose used three times a week (TIW) in alternate days in monotherapy. 29 days of treatment. Subcutaneous injection.
  Arms: Interferon α-5
Drug: Interferon-α5 plus Interferon-α 2b — Interferon-α5 plus Interferon-α 2b. 1.5 MIU each, or safe dose used TIW in alternate days in combined therapy. 29 days of treatment. Subcutaneous injection.
  Arms: Interferon α-5 plus Interferon α-2b
Drug: Interferon α-2b (INTRON® A) — 3 million IU TIW in alternate days in monotherapy. 29 days of treatment. Subcutaneous injection.
  Arms: Interferon α-2b (INTRON® A)

SUMMARY:
The general aim of this study is to determine if 3 MIU of IFN-α5 in monotherapy, and 1,5 MIU of IFN-α5 combined with 1,5 MIU of IFN- α2b, are safe dose levels as well as to investigate the antiviral efficacy and pharmacodynamics (PD) of such doses and drugs in treatment-experienced HCV patients with genotype 1 chronic infection, after 29 days of treatment. It is also intended to determine pharmacokinetics (PK) of the safe dose achieved of IFN-α5 in monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old,
2. With chronic hepatitis C (CHC) infection diagnosed by seropositivity for anti-HCV antibodies or detectable HCV-RNA, at least 6 months prior to screening.
3. Patients with CHC infection of genotype 1 (1a, 1b or mixed 1a/1b)
4. Defined as relapsers: those CHC patients who had achieved virologic response (HCV-RNA non detectable) at any time during the standard care of treatment for CHC with IFN-α2 or PegIFN-α2 + ribavirin, and maintained it trough the end of treatment at week 48 weeks, but HCV-RNA detection occurs before 6 months post-treatment.
5. In whom liver cirrhosis has been ruled out through fibro-scan or liver biopsy within 24 months prior to study enrolment.
6. With a serum HCV viral load ≥ 100.000 IU/mL at screening
7. With alanine-aminotransferase (ALT) and aspartate-aminotransferase (AST) serum measurements at screening less than 5 times of their upper limits of normal (ULN)
8. With a body mass index (BMI) of at least 18 kg/m2, but not exceeding 36 kg/m2.
9. For female subjects with childbearing potential: use of a known highly effective method of birth control
10. For male subjects with partners of child bearing potential: use of appropriate contraceptive methods.
11. Is able to effectively communicate with the investigator and other testing center personnel.
12. Is able to participate and willing to give written informed consent and comply with the study restrictions.

Exclusion Criteria(principal):

1. Hepatitis C infection of genotype 2, 3 or 4 or any mixed genotype (1/2, 1/3 and 1/4).
2. A positive ELISA for HIV-1 or HIV-2.
3. Hepatitis B virus (HBV) infection based on the presence of HBsAg.
4. Hepatitis A virus (HAV) infection based on the presence of antiHAV-IgM. (AM 4)Criteria deleted
5. Decompensated liver disease, or history of decompensated liver disease.
6. History or other evidence of a medical condition associated with decompensated renal, immunologically mediated, chronic pulmonary, cardiac, thyroid, severe retinopathy, severe psychiatric, organ transplantation, cancer, seizure disorder or pancreatitis diseases.
7. An active or suspected malignancy or history of malignancy within the last five years.
8. Patients with a documented drug and alcohol addiction free history of at least 12 months who are, in the opinion of the investigator unlikely to relapse, may be enrolled in the study.
9. Positive results for drug abuse at screening.Occasional use of cannabis previously to randomization is not an exclusion criteria -under investigator team criteria-. The patient should be advised of abstinence during the trial (AM 6)
10. Haemoglobin <12.0g/dL for women, and <13.0g/dL for men at screening.
11. White blood cell count <2000 cells/mm3 at screening.
12. Absolute neutrophil count <1500 cells/mm3 at screening.
13. Platelet count <100.000 cells/mm3 at screening.
14. ALT and AST levels ≥ 5 xULN at screening.
15. Prothrombin time INR prolonged to 1.5xULN at screening.
16. TSH an T4 outside normal limits and not adequately controlled thyroid function at screening.
17. Poorly controlled diabetes mellitus as evidenced by HbA1c >7.5% at screening.
18. Alfa-fetoprotein value >100ng/mL at screening.
19. Total bilirubin >1.5xULN with ratio of direct/indirect >1, at screening unless predominantly conjugated and reflecting Gilbert's disease
20. Estimated creatinine clearance of 30 mL/minute or less at screening.
21. Women who are confirmed to be pregnant
22. People with known hypersensitivity to any ingredient of the investigational agents
23. Patients who are at risk of bleeding.
24. Haemoglobinopathy
25. Screening ECG QTc value ≥ 450ms and/or clinically significant ECG findings.
26. History of clinically significant drug allergies.
27. Participation in a clinical study with an investigational drug, biologic, or device within 3 months prior to anticipated dose administration.
28. Any chronic viral (including HSV), bacterial, mycobacterial, fungal, parasitic, or protozoal infection.
29. Requirement for chronic systemic corticosteroids.
30. Receiving systemic antivirals, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safe dose level | 29 days of treatment
  PRIMARY ENDPOINTS OF PHASE I
  * To determine if 3 MIU of IFN-α5 are well tolerated and if not, to find a safe dose level for IFN-α5.
  * To determine if 1.5 MIU of IFN-α5 in combination with 1.5 MIU of IFN-α2b (IFN-α5 + IFN-α2b) are well tolerated and if not, to find a safe dose level for the combination of IFN-α5 and IFN-α2b.
  PRIMARY ENDPOINTS OF PHASE II
  * To analyze IFN-α5 preliminary antiviral efficacy at the dose of 3 MIU, or the safe dose level identified in Phase I.
  * Primary safety endpoints: Occurrence of AE (classified into mild, moderate and severe)

SECONDARY OUTCOMES:
pharmacodynamic and pharmacokinetic parameters | 29 days of treatment
  SECONDARY ENDPOINTS OF PHASE I
  * To obtain pharmacokinetic parameters of IFN-α5 in monotherapy after single and multiple dose administration
  * To obtain pharmacodynamic parameters of IFN-α5 in monotherapy and in combination with IFN-α2b
  SECONDARY ENDPOINTS OF PHASE II
  * To analyze IFN-α5 + IFN-α2b preliminary antiviral efficacy and comparison between IFN-α5 in monotherapy, IFN-α5 + IFN-α2b and IFN-α2b in monotherapy.
  * To obtain pharmacodynamic parameters after treatment with IFN-α5, IFN-α5 + IFN-α2b or IFN-α2b.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Prieto, MD, PhD, Principal Investigator — Clínica Universidad de Navarra. Spain
Locations (15):
- Spain (15):
  - Centre 013, A Coruña
  - Centre 004, Barcelona
  - Centre 005, Barcelona
  - Centre 008, Barcelona
  - Centre 011, Barcelona
  - Centre 014, Granada
  - Centre 015, León
  - Centre 002, Madrid
  - Centre 003, Madrid
  - Centre 006, Madrid
  - Centre 009, Madrid
  - Centre 016, Madrid
  - Centre 001, Pamplona
  - Centre 012, Santander
  - Centre 010, Seville